CLINICAL TRIAL: NCT06099808
Title: Randomized Evaluation of Audit and Feedback Intervention to Promote Pharmacist Heart Failure Medication Titration in Veterans Affairs Sierra Pacific Network
Brief Title: Veterans Affairs Pharmacist Heart Failure Medication Titration Project 1
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul A. Heidenreich, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 72662
Record Dates: First submitted 2023-10-18; First posted 2023-10-25 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: Pharmacist; Medication therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Audit and Feedback (AF) (Experimental): Pharmacists randomized to audit and feedback will receive a monthly email containing information including their total medication titration encounters over a 3 month period, as well as the site and VISN level for comparison. The audit and feedback email will also contain rates of medical therapy and percentage of patients on >50% of the target dose of medical therapy stratified by site, VISN and national. This data will be obtained from VHA national HF dashboard. Pharmacists in AF will also receive invitations to monthly educational sessions and access to shared resources on HF medication management.
  Interventions: Other: Audit and Feedback Emails; Other: Educational Resources
- Audit and Feedback with Patient Specific Targets (AF+) (Experimental): Pharmacists randomized to the AF+ group will receive the audit and feedback intervention described above with the addition of a list of 5-7 HF patients who are potentially eligible for pharmacist HF medication titration. These patients will be identified using the VHA national HF dashboard.
  Interventions: Other: Audit and Feedback Emails; Other: Patient Specific Targets; Other: Educational Resources
- Usual Care (Active Comparator): Pharmacists randomized to the usual care arm will have access to monthly educational sessions and to shared resources on HF medication management. They will receive no additional feedback.
  Interventions: Other: Educational Resources

INTERVENTIONS:
Other: Audit and Feedback Emails — Monthly email containing information including their total medication titration encounters over a 3 month period, as well as the site and VISN level for comparison. This will include rates of GDMT utilization and percentage of patients on >50% of the target dose of GDMT stratified by site, VISN and national. This data will be obtained from VHA national HF dashboard.
  Arms: Audit and Feedback (AF); Audit and Feedback with Patient Specific Targets (AF+)
Other: Patient Specific Targets — Monthly emails include a list of 5-7 HF patients who are potentially eligible for pharmacist HF medication titration. This data will be obtained from VHA national HF dashboard.
  Arms: Audit and Feedback with Patient Specific Targets (AF+)
Other: Educational Resources — Monthly educational webinars on pharmacist HF management and access to material and protocols on HF medication management.

SUMMARY:
This is a randomized quality improvement project to evaluate the impact of an audit and feedback intervention to motivate pharmacists to provide heart failure (HF) medication management to patients in the Veterans Health Administration (VHA) Sierra Pacific region (VISN 21). The results of this project could provide guidance for how to successfully scale a pharmacist-based HF remote management program in the VHA more broadly.

Pharmacists providing clinical care as part of Patient Aligned Care Team (PACT) within VHA VISN 21 will be included. Pharmacists will be randomized to one of 3 arms in a 1:1:2 ratio: (1) monthly audit and feedback of HF medication titration activities (AF) vs. (2) educational resources and monthly notification of HF medication titration actions in addition to a list of potential patients for HF optimization (AF+) vs. (3) usual care without audit and feedback (UC). Pharmacists across all three arms will be given access to shared educational resources on HF pharmacist care and educational webinars. Six months after the intervention, rates of pharmacist HF medication titration encounters will be compared among the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical pharmacists in the Veterans Health Administration that provide Patient Aligned Care Team (PACT) care in VA Sierra Pacific Network (VISN 21)

Exclusion Criteria:

* Excluded per pharmacist supervisor decision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of monthly heart failure medication adjustment encounters | 2 months post-randomization to 6 months post-randomization
  Encounters in which pharmacist adjusted heart failure medications

SECONDARY OUTCOMES:
Percentage of heart failure patients with medication management by pharmacist | Within 6 months post-randomization
  For each pharmacist, will calculate the percentage of patients with heart failure in their panel that receive medication adjustments from pharmacist
Number of new patients with pharmacist HF management | Within 6 months post-randomization
  For each pharmacist, will calculate the number of patients with heart failure in their panel that receive care from pharmacist that were not receiving care prior to randomization
Guideline medical therapy score | At 6 months post randomization
  Composite score of heart failure medical therapy among patients with heart failure for patients within each pharmacists panel
Beta-blocker therapy | At 6 months post randomization
  Percentage of patients with heart failure with reduced ejection fraction in each pharmacist panel that are treated with beta-blocker therapy
Renin-angiotensin system inhibitor (RASI) therapy | At 6 months post randomization
  Percentage of patients with heart failure with reduced ejection fraction in each pharmacist panel that are treated with RASI therapy
Angiotensin receptor neprilysin inhibitor (ARNI) therapy | At 6 months post randomization
  Percentage of patients with heart failure with reduced ejection fraction in each pharmacist panel that are treated with ARNI therapy
Mineralocorticoid receptor antagonist (MRA) therapy | At 6 months post randomization
  Percentage of patients with heart failure in each pharmacist panel that are treated with MRA therapy
Sodium-Glucose Cotransporter-2 Inhibitor (SGLT2i) therapy | At 6 months post randomization
  Percentage of patients with heart failure in each pharmacist panel that are treated with SGLT2i therapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Heidenreich, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Palo Alto Veteran's Affairs Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No